CLINICAL TRIAL: NCT02813317
Title: Optimizing the Care Pathways of Patients Treated for Operable Breast Cancer
Brief Title: Optimizing the Care Pathways of Patients Treated for Operable Breast.
Acronym: OPTIsoins01
Status: Completed | Type: Observational
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Other Study IDs: IC 2014-11
Record Dates: First submitted 2016-01-06; First posted 2016-06-27 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Surgery
Keywords: Surgery; Breast cancer; Quality of life; Care pathway; Economic evaluation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective, multicenter, observational study aims to explore a comprehensive approach to the care of early breast cancer patients in a regional health territory (including 1.5 million women and characterized by a breast cancer incidence and mortality higher than national ranges), incorporating all healthcare actors inside and outside the hospital.

DETAILED DESCRIPTION:
The treatment course of a breast cancer patient includes a hospital stay, home health care that requires outpatient services, supportive care and a follow-up course. Outpatient surgery and home hospitalization units are two innovative organizational technologies that are strongly recommended because of their putative positive medico-economic impact; however, these structures are poorly studied in terms of quality of care and patient satisfaction. Regional implementation of these innovations is heterogeneous, thus allowing a comparative study.

This prospective, multicenter, observational study aims to explore a comprehensive approach to the care of early breast cancer patients in a regional health territory (including 1.5 million women and characterized by a breast cancer incidence and mortality higher than national ranges), incorporating all healthcare actors inside and outside the hospital.

This study will be conducted in academic centers, general hospitals and private centers. In the different participating centers, the implemented care steps are different and may include outpatient surgery, home hospitalization, a one-stop breast clinic visit, care by an oncology pivot nurse and/or screening for supportive care. Outpatient surgery and home hospitalization in particular are two health technologies that are validated by the French National Authority for Health but used differently in different centers.

The primary objective is to examine the economic and financial measurements of the different care pathways of early breast cancer patients to compare the economic burden of outpatient surgery and home hospitalization with the conventional care pathway.

The secondary objectives are:

Assessing patient satisfaction and needs for supportive care. Evaluating the structures and organizations. Evaluating the tool exchanges between the actors over the treatment course.

All parameters related to the patient and to disease characteristics, determinants and management characteristics within and outside the center within one year will be collected and centralized in the study database. The patients' course of care will be divided into five stages: preadmission, hospitalization, the postoperative period (+ 1 month), adjuvant treatments and one-year follow-up. Care pathways will be identified, described and analyzed to meet the primary objective and the secondary objectives.

After analyzing these care pathways, we will propose solutions for optimizing hospital and nonhospital care, thereby building efficient connections among the hospital, home health care, district nurse networks, medical and social sectors, and occupational reintegration.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent.
2. Patients aged ≥18 years.
3. Previously untreated, operable breast cancer
4. Affiliation with the social security system (or a similar coverage)
5. Patient living in one of these french department : "Hauts-de-Seine (92)", "les Yvelines (78)", or "le Val d'Oise (95)".
6. Female gender.

Exclusion Criteria:

1. Previous history of breast cancer.
2. Metastatic, locally advanced, or inflammatory breast cancer, as defined by the AJCC (American Joint Committee on Cancer, 7th Edition).
3. Any prior treatment for primary breast cancer.
4. Patient with any psychological, sociological or geographical condition potentially hampering compliance with the study follow-up schedule.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Previously untreated, operable breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 617 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Care pathways description of early breast cancer patients. | Up to one year after patient registration
  Care pathways will be characterized by the sequence of different care steps. Care steps may include : outpatient surgery, home hospitalization, a one-stop breast clinic visit, care by an oncology pivot nurse and/or screening for supportive care.
Overall cost measurements of the different care pathways. | Up to one year after patient registration
  Evaluating the overall costs of the pathway care (health care and supportive care consumption) at one year for the different perspectives.
Overall cost measurements of the different care pathways for health insurance | Up to one year after patient registration
  Evaluating the indirect costs of health insurance
Overall cost measurements of the different care pathways for the patient | Up to one year after patient registration
  Evaluating the out-of-pocket health expenses for breast cancer during the first year post diagnosis (direct and indirect costs).

SECONDARY OUTCOMES:
Patient satisfaction evaluation | Up to one year after patient registration.
  Patient satisfaction will be assessed at different time points using the OUT-PATSAT35 questionnaire validated in French.
Supportive care needs assessement | Up to one year after patient registration
  The patient's needs for supportive care will be assessed using the Supportive Care Needs Survey - Breast Cancer module (SCNS-BR8) validated in French.
Supportive care needs assessement | Up to one year after patient registration
  The patient's needs for supportive care will be assessed using the Supportive Care Needs Survey Short Form (SCNS-SF34) validated in French.
Breast cancer impact on patient's professional activity | Up to one year after patient registration.
  Evaluating patient return to work : Existence of an occupational reintegration or not.
Breast cancer impact on patient's professional activity | Up to one year after patient registration.
  Evaluating patient return to work : Date of return to work
Breast cancer impact on patient's professional activity | Up to one year after patient registration.
  Evaluating patient return to work : Organization of working time description
Breast cancer impact on patient's professional activity | Up to one year after patient registration.
  Evaluating patient return to work : Number of days out of work
Structures and organizations interactions description | Up to one year after patient registration
  Identification of health care actors inside and outside the hospital
Structures and organizations interactions description | Up to one year after patient registration
  identification of the interactions between the organizations (e.g., identification, shared tools, resource sharing and nurse training).
Structures and organizations interactions description | Up to one year after patient registration
  Regular practitioners questionnaires

OTHER OUTCOMES:
Care pathways suggestion for a regional health territory. | Through study completion (within one year after the last patient follow-up)
  After analyzing these care pathways, we will propose solutions for optimizing hospital and nonhospital care, thereby building efficient connections among the hospital, home health care, district nurse networks, medical and social sectors, and occupational reintegration.

CONTACTS AND LOCATIONS:
Overall Officials: Roman ROUZIER, Pr, Study Director — Institut Curie; Delphine HEQUET, MD PhD, Study Director — Institut Curie
Locations (9):
- France (9):
  - Victor Dupouy Hospital, Argenteuil
  - Antoine Béclère Hospital, Clamart
  - Louis Mourier Hospital, Colombes
  - André Mignot Hospital - Versailles, Le Chesnay
  - Institut Curie, Paris
  - Bichat Beaujon University Hospital, Paris
  - Poissy Interegional Hospital Center, Poissy
  - René Dubos Hospital, Pontoise
  - Institut Curie - René Huguenin Hospital, Saint-Cloud

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arfi A, Baffert S, Soilly AL, Huchon C, Reyal F, Asselain B, Neffati S, Rouzier R, Hequet D. Determinants of return at work of breast cancer patients: results from the OPTISOINS01 French prospective study. BMJ Open. 2018 May 18;8(5):e020276. doi: 10.1136/bmjopen-2017-020276. PMID 29776920